CLINICAL TRIAL: NCT05832931
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Dose-Titrated PLS240 in the Treatment of Secondary Hyperparathyroidism in Individuals With End Stage Kidney Disease on Hemodialysis (PATH-1) With an Open-Label Extension
Brief Title: Parathyroid Hormone (PTH) Attenuation Trial in Hemodialysis-1
Acronym: PATH-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pathalys Pharma (Industry)
Collaborators: Launch Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PP3002; 2023-504338-24 (EudraCT Number)
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Secondary Hyperparathyroidism; End-stage Kidney Disease (ESKD)
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Double-Blind Phase PLS240 (Experimental)
  Interventions: Drug: PLS240
- Double-Blind Phase Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Open-Label Extension Phase PLS240 (Experimental): After completion of the Double-Blind Phase, all participants will have the opportunity to enroll in the 26 week Open-Label extension, where they will receive PLS240.
  Interventions: Drug: Open-Label Extension PLS240

INTERVENTIONS:
Drug: PLS240 — Participants will receive intravenous (IV) PLS240 three times per week for 27 weeks.
  Arms: Double-Blind Phase PLS240
Drug: Placebo — Participants will receive intravenous (IV) placebo, containing no active drug, three times per week for 27 weeks.
  Arms: Double-Blind Phase Placebo
Drug: Open-Label Extension PLS240 — Participants will receive intravenous (IV) PLS240 three times per week for a maximum of 26 weeks.
  Arms: Open-Label Extension Phase PLS240

SUMMARY:
This study is to evaluate the efficacy and safety of PLS240 in patients with hemodialysis-dependent end stage kidney disease (ESKD) and secondary hyperparathyroidism (SHPT). The study consists of two phases. First, a placebo-controlled, double-blind phase where patients will be randomly assigned to either receive dose-titrated PLS240 or matching placebo for 27 weeks. After the completion of the double-blind phase, patients will be eligible to enroll in the open-label extension phase, where they will receive dose-titrated PLS240 for an additional 26 weeks. Throughout the duration of the study, patients will be expected to attend multiple study visits where an investigator will collect blood, preform electrocardiograms (ECGs) and physical exams, and further assess the safety and efficacy of PLS240.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 80 years at time of informed consent.
2. Prescribed hemodialysis for 3 times per week and on therapy for at least 3 months and has a delivered Kt/V≥1.2 within 4 weeks prior to signing the ICF.
3. Pre-dialysis central laboratory iPTH must be ≥400 pg/mL on at least two assessments performed at 2 visits, at least 1 week apart during the Active Screening period. iPTH may be tested up to 4 times.

   at least performed at least a week after the previous iPTH.
4. Pre-dialysis central laboratory cCa must be ≥8.3 mg/dL on at least one assessment performed during the Active Screening period. cCa may be tested up to 3 times during the Active Screening period.
5. Dialysate calcium concentration ≥2.5 mEq/L (1.25 mmol/L) and stable for at least 4 weeks prior to signing the ICF.
6. Participants receiving active Vitamin D sterols (e.g., doxercalciferol or calcitriol) to manage SHPT must be on a stable dose (e.g., maximum dose change ≤50%), in the opinion of the investigator or sub-investigator, within the 2 months prior to signing the ICF, remain stable, as defined as no increase in dose, through the screening period, and be expected to maintain a stable dose, as defined as no increase in dose, for the duration of the study.
7. Participants receiving phosphate binders must be on a stable dose (e.g., maximum dose change ≤50%), in the opinion of the investigator or sub-investigator, within the 2 months prior to signing the ICF, remain stable through the screening period, and be expected to maintain stable dose for the duration of the study.
8. Participants receiving calcium supplements must be on a stable dose (e.g., maximum dose change ≤50%), in the opinion of the investigator or sub-investigator, within the 2 months prior to signing the ICF and remain stable through the screening period.
9. Female participants who are post-menopausal ('post-menopausal' women have had no menses for the previous year and are over the age of 50 years), or surgically sterilized, or have a medical condition that prevents pregnancy, or commit to remain abstinent during the study and for 2 weeks after the last dose of the investigational product (IP), or are willing to use highly effective contraception during the study and for 2 weeks after the last dose of IP. Women of child-bearing potential must have a negative serum pregnancy test during the screening period.
10. Male participants who are willing to use highly effective contraception when sexually active and will not donate sperm during the treatment phase and for 2 weeks after the last dose of IP.
11. Voluntarily given written informed consent to participate in this study.
12. Agrees to not participate in another study of an investigational agent during the study

    To be eligible for inclusion into the Open-Label Extension Phase of the study, participants must fulfill the additional following criteria at the time of entry into the Open-Label Extension Phase:
13. Have successfully completed the course of treatment and final safety follow-up visit of the Double-Blind Phase.
14. Voluntarily given written informed consent to participate in the Open-Label Extension Phase of the study.
15. Prescribed hemodialysis for 3 times per week. 16. Continue to meet Inclusion Criteria 9, 10, and 12.

Exclusion Criteria:

1. Diagnosis of primary hyperparathyroidism.
2. Pre-dialysis central laboratory Active Screening iPTH >1500 pg/mL on two or more occasions. iPTH may be tested up to 4 times during the Active Screening period.
3. History of parathyroid intervention including parathyroidectomy (PTx) and percutaneous ethanol injection therapy (PEIT) within 26 weeks before signing the ICF.
4. Treatment with any prohibited medication as defined in Section 8.3.1.
5. Anticipated or scheduled parathyroidectomy during the study period.
6. Planned living-related or living-unrelated kidney transplant during the study period.
7. Change in mode of dialysis (e.g., from hemodialysis to hemodiafiltration, peritoneal dialysis to hemodialysis, at home to in center dialysis), dialysate Ca concentration, or prescribed dialysis treatment time within 4 weeks before signing the ICF.
8. Noncompliant with hemodialysis (i.e., missing more than 2 dialysis sessions within 8 weeks prior to signing the ICF, unless absence is due to hospitalization or dialysis-access procedures).
9. Clinically significant abnormalities on screening laboratory tests (may repeat abnormal laboratory tests) according to the Investigator including but not limited to the following:

   1. Serum albumin ≤3.0 g/dL
   2. Serum magnesium <1.5 mg/dL
   3. Serum P >8.0 mg/dL
   4. Hemoglobin <8.5 g/dL
   5. Platelet count <100,000 x106/L
   6. Serum transaminase (alanine transaminase [ALT] or serum glutamic pyruvic transaminase [SGPT], alanine transaminase [AST] or serum glutamic oxaloacetic transaminase [SGOT]) ≥2.5 times the upper limit of normal (ULN) during Active Screening.
10. Diagnosed with an unstable medical condition, defined as having been hospitalized, other than for dialysis vascular access intervention, within 30 days prior to signing the TCF, or otherwise unstable in the judgment of the investigator.
11. History of malignancy within the last 2 years prior to signing the ICF (except squamous or basal cell skin cancers, or cervical carcinoma in situ).
12. Recent history (within 4 weeks prior to signing the ICF) of angina pectoris with symptoms that occur at rest or minimal activity. Chest pain on dialysis (within 8 weeks prior to signing the ICF) unless evaluated by a cardiologist with documentation that the chest pain is not due to cardiac ischemia.
13. History of New York Heart Association (NYHA) Functional Class 3 or 4 heart failure.
14. History of myocardial infarction, coronary angioplasty, or coronary arterial bypass grafting within the past 4 months prior to signing the ICF.
15. Stroke (cerebral infarction or cerebral hemorrhage) within 6 months prior to signing the ICF.
16. Participant is receiving treatment for a seizure disorder or has a history of a seizure within 12 weeks prior to signing the ICF.
17. Poorly controlled diabetes mellitus, in the judgment of the investigator or sub-investigator.
18. Poorly controlled hypertension (defined as post-dialysis [seated if available] systolic pressure >180 mmHg or diastolic pressure >110 mmHg) at 2 or more dialysis sessions during the 2 weeks prior to signing the ICF.
19. Enrolled in other invasive investigational device or investigational drug trials, within at least 30 days prior to signing the ICF or are receiving other investigational agents (experimental dialysis machines are acceptable).
20. History of symptomatic ventricular dysrhythmias or Torsade de Pointes.
21. History of or family history of long QT syndrome.
22. QTcF >500 msec on screening ECG.
23. Pregnant or breast feeding.
24. Prior exposure or hypersensitivity to PLS240 or any of its components.
25. Current, recent, or suspected infection with SARS-CoV-2/COVID-19 within 4 weeks prior to signing the ICF.
26. In the opinion of the investigator, any disorder that would interfere with understanding and giving informed consent, or compliance with protocol requirements.

    Participants must be excluded from the Open-Label Extension Phase of the study, in case of the following at the time of entry into the Open-Label Extension Phase:
27. In the opinion of the investigator, continuation into the Open-Label Extension Phase is not considered safe and/or feasible.
28. Continues to meet Exclusion Criterion #5.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Double-Blind Phase: Proportion of PLS240 treated participants compared to placebo treated participants with a ≥30% decrease in mean iPTH | each visit from screening through week 27
  This measurement will be calculated based on the Efficacy Assessment Period (Weeks 22 - 27) relative to the mean baseline iPTH (all Active Screening and predose Day 1 iPTH values).
Open-Label Phase: Proportion of participants with a corrected serum calcium (cCa) <7.5 mg/dL | up to week 28
Open-Label Phase: Proportion of participants with a corrected serum calcium (cCa) <8.3 mg/dL | up to week 28
Open-Label Phase: Number of Adverse Events (AEs) | up to week 28
Open-Label Phase: Number of Serious Adverse Events (SAEs) | up to week 28

CONTACTS AND LOCATIONS:
Locations (68):
- United States (49):
  - Site Number: USA016-1, Pine Bluff, Arkansas
  - Site Number: USA032-1, Anaheim, California
  - Site Number: USA031-1, Beverly Hills, California
  - Site Number: USA020-1, Fairfield, California
  - Site Number: USA023-1, Fullerton, California
  - Site Number: USA030-1, Glendale, California
  - Site Number: USA045-1, Oxnard, California
  - Site Number: USA046-1, Riverside, California
  - Site Number: USA035-1, Salinas, California
  - Site Number: USA001-1, San Diego, California
  - Site Number: USA021-1, San Diego, California
  - Site Number: USA019-1, San Dimas, California
  - Site Number: USA036-1, Whittier, California
  - Site Number: USA018-1, Denver, Colorado
  - Site Number: USA003-1, Lone Tree, Colorado
  - Site Number: USA009-1, Hartford, Connecticut
  - Site Number: USA042-1, Coral Gables, Florida
  - Site Number: USA055-1, Coral Gables, Florida
  - Site Number: USA034-1, Hollywood, Florida
  - Site Number: USA053-1, Atlanta, Georgia
  - Site Number: USA013-1, Dalton, Georgia
  - Site Number: USA027-1, Boise, Idaho
  - Site Number: USA007-1, Shelbyville, Indiana
  - Site Number: USA026-1, Baton Rouge, Louisiana
  - Site Number: USA015-1, Columbus, Mississippi
  - Site Number: USA028-1, Oxford, Mississippi
  - Site Number: USA022-1, Kansas City, Missouri
  - Site Number: USA017-1, Las Vegas, Nevada
  - Site Number: USA010-1, Jersey City, New Jersey
  - Site Number: USA008-1, Gallup, New Mexico
  - Site Number: USA039-1, Manhasset, New York
  - Site Number: USA011-1, The Bronx, New York
  - Site Number: USA052-1, Charlotte, North Carolina
  - Site Number: USA043-1, Greenville, North Carolina
  - Site Number: USA033-1, Winston-Salem, North Carolina
  - Site Number: USA040-1, Spartanburg, South Carolina
  - Site Number: USA049-1, Knoxville, Tennessee
  - Site Number: USA037-1, Arlington, Texas
  - Site Number: USA024-1, Austin, Texas
  - Site Number: USA056-1, Fort Worth, Texas
  - Site Number: USA014-1, Houston, Texas
  - Site Number: USA012-1, Houston, Texas
  - Site Number: USA025-1, McAllen, Texas
  - Site Number: USA029-1, San Antonio, Texas
  - Site Number: USA005-1, San Antonio, Texas
  - Site Number: USA004-1, San Antonio, Texas
  - Site Number: USA002-1, The Woodlands, Texas
  - Site Number: USA006-1, Norfolk, Virginia
  - Site Number: USA050-1, Wauwatosa, Wisconsin
- Bulgaria (4):
  - Site Number: BGR003-1, Sofia, Sofia-Grad
  - Site Number: BGR004-1, Sofia, Sofia-Grad
  - Site Number: BGR002-1, Blagoevgrad
  - Site Number: BGR001-1, Plovdiv
- Poland (2):
  - Site Number: POL005-1, Oleśnica, Lower Silesian Voivodeship
  - Site Number: POL002-1, Żyrardów, Masovian Voivodeship
- Portugal (3):
  - Site Number: PRT003-1, Portimão, Faro District
  - Site Number: PRT001-1, Carregado, Lisbon District
  - Site Number: PRT002-1, Forte Da Casa, Lisbon District
- Serbia (4):
  - Site Number: SRB001-1, Belgrade
  - Site Number: SRB003-1, Kragujevac
  - Site Number: SRB005-1, Novi Sad
  - Site Number: SRB002-1, Zaječar
- Spain (6):
  - Site Number: ESP001-1, Lleida
  - Site Number: ESP004-1, Madrid
  - Site Number: ESP005-1, Madrid
  - Site Number: ESP003-1, Pamplona
  - Site Number: ESP006-1, Seville
  - Site Number: ESP002-1, Valencia

IPD SHARING:
Plan to Share IPD: No